CLINICAL TRIAL: NCT07136727
Title: The Impact of Multimodal Digital Fusion AI-Assisted Decision Support System-Based Comprehensive Management on Clinical Outcomes in County-Level Patients With Comorbid Cancer:A Prospective Non-randomized Controlled Interventional Study.
Brief Title: AI-Assisted Comprehensive Management for Cancer Patients With Comorbidities (GCOG-CG001)
Acronym: GCOG-CG001
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCOG-CG001
Record Dates: First submitted 2025-08-09; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Oncological Comorbidities (e. g. Hypertension, Diabetes, Malnutrition)
Keywords: Malignant neoplasm; Comorbidity; Artificial intelligence
MeSH Terms: conditions — Diabetes Mellitus; Malnutrition; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI management unit (Experimental): For patients with comorbid pulmonary malignancies who have been included, the registration process is guided by the management platform. Researchers will use digital management throughout The platform carries out screening assessment and Comprehensive Evaluation of nutrition, exercise, psychology and symptoms of the subjects, and the system will be combined with the patient's disease and treatment Information, intelligent management of the whole project. The clinician can review the protocol in the light of the patient's disease status and give the full management instructions Case to patient side.
  Interventions: Other: AI-assisted comprehensive management system
- Standard Clinical Management (No Intervention): Patients who are not willing to accept the whole program will only be followed up, and will receive standard clinical management without AI-assisted digital platform support. Patients will receive conventional treatment. In the data analysis phase, subjects were stratified to explore the feasibility and effectiveness of digital whole-course management in patients with oncological comorbidities.

INTERVENTIONS:
Other: AI-assisted comprehensive management system — Precision Risk Stratification and personalized treatment recommendation through AI models may improve the suitability of treatment regimens and thus reduce the incidence of antineoplastic therapy-related adverse effects (e.g. , reduction of chemotherapy toxicity through nutritional intervention) , and improve the efficacy of chemotherapy, and prolonged progression-free survival (PFS) and overall survival (OS)
  Arms: AI management unit

SUMMARY:
Combined with the digital whole process management data pool, a multi-modal data fusion framework is developed, and an AI model is established to realize risk stratification and personalized treatment Recommendation and dynamic prognosis prediction; validation of whole-process management based on multimodal digital fusion AI-aided decision support system through prospective non-randomized controlled interventional study The effect on survival, complication control and utilization of medical resources in patients with comorbid malignant tumors.

DETAILED DESCRIPTION:
The title of this study is"The Impact of Multimodal Digital Fusion AI-Assisted Decision Support System-Based Comprehensive Management on Clinical Outcomes in County-Level Patients with Comorbid Cancer: A prospective non-randomized controlled interventional study", to evaluate the impact of full-course management based on a multimodal digital fusion AI-assisted decision support system on the clinical outcomes of county-level oncologic comorbid patients through a prospective non-randomized controlled interventional study. The study plans to enroll 5,000 patients with pathologically confirmed malignancies and at least one comorbid condition (diabetes, hypertension, etc.) , in the first stage, the epidemiological characteristics of co-morbidity and its impact on prognosis, treatment response and quality of life were analyzed In the second phase, patients with comorbid pulmonary malignancies were selected to compare the clinical effects of the voluntary whole-process management group (including personalized intervention such as nutritional screening and dynamic monitoring) and the conventional treatment group, the third stage integrates multi-center Electronic Medical Records, genomic data, wearable device monitoring and other multi-modal data to construct an AI decision-making system, developing risk stratification, personalized treatment recommendation, and dynamic prognostic prediction models, finally, the differences in core indicators such as survival rate (PFS, OS) , complication control and medical resource efficiency between AI-assisted management and traditional mode were compared. This study realizes the integrated intervention of in-hospital and out-of-hospital through digital whole-process management, which is expected to provide an AI-driven precise decision support paradigm for primary medical institutions and improve the efficiency of comprehensive management of tumor comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite diagnosis of malignancy by histopathology and/or cytology;
* Age ≥18 years;
* There is no gender limit
* Plan to receive antineoplastic therapy within 2 weeks or are receiving standard antineoplastic care (surgery, radiation, chemotherapy, or targeted therapy) ;
* Conscious and able to answer questions and use electronic devices autonomously;
* Patients were able to understand the study and voluntarily sign an informed consent form;

Exclusion Criteria:

* Having severe mental or cognitive impairments that prevent them from understanding the content of the study or implementing the programme;
* With severe heart disease, acute respiratory failure, liver kidney failure and other critical illness;
* Women during pregnancy or lactation；
* Have participated in other interventional studies in the past 1 month or are currently participating;
* Patients with ECOG ≥ 3 that do not respond to treatment;
* Patients with an expected survival of < 3 months that do not respond to treatment;
* Cases deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Progression-free survival (PFS) : the time from randomization (or study enrollment) to the observation of disease progression or the occurrence of death from any cause. This period was assessed every 6-8 weeks using RECIST 1.1 criteria.
Overall survival (OS） | 24 months
  Overall survival (OS） : the time from study enrollment to death from any cause from any cause, every 3 months during treatment, and every 3 months after the end of treatment. The patients were followed up at 6 months and the cause of death was recorded.

SECONDARY OUTCOMES:
Comorbidity control rate. | 24 months
  Comorbidity control rate: the proportion of comorbidities achieving guideline-recommended control targets during the study period; stratified criteria should be established based on specific comorbidity types.
Quality of life(QLQ-C30). | 24 months
  Quality of life: changes in scores at baseline, on-treatment, and follow-up were assessed using the European Organisation for Research and Treatment of Cancer QLQ-C30 scale, between-group differences
Medical resource consumption index. | 24 months
  Medical resource consumption index: Comparing DRG-adjusted medical resource consumption indices between two groups.
Adherence to AI system interventions. | 24 months
  Adherence to AI Interventions:
  1. In-Hospital Rate - Percentage of inpatients completing AI-recommended actions (e.g., nutritional screening, real-time monitoring).
  2. Out-of-Hospital Completion Rate: Percentage of discharged/outpatients adhering to AI-guided care (e.g., telehealth, wearable data tracking).
  Enables precise evaluation of AI-driven care across clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shen Wei Shen, MD, Doctor of Medicine, Study Chair — First Affiliated Hospital of Xinjiang Medical University
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No
Data security and privacy protection measures.

REFERENCES:
- [Background] Stairmand J, Signal L, Sarfati D, Jackson C, Batten L, Holdaway M, Cunningham C. Consideration of comorbidity in treatment decision making in multidisciplinary cancer team meetings: a systematic review. Ann Oncol. 2015 Jul;26(7):1325-32. doi: 10.1093/annonc/mdv025. Epub 2015 Jan 20. PMID 25605751
- [Background] Ding R, Zhu D, He P, Ma Y, Chen Z, Shi X. Comorbidity in lung cancer patients and its association with medical service cost and treatment choice in China. BMC Cancer. 2020 Mar 24;20(1):250. doi: 10.1186/s12885-020-06759-8. PMID 32209058
- [Background] Chao C, Page JH, Yang SJ, Rodriguez R, Huynh J, Chia VM. History of chronic comorbidity and risk of chemotherapy-induced febrile neutropenia in cancer patients not receiving G-CSF prophylaxis. Ann Oncol. 2014 Sep;25(9):1821-1829. doi: 10.1093/annonc/mdu203. Epub 2014 Jun 10. PMID 24915871
- [Background] Sogaard M, Thomsen RW, Bossen KS, Sorensen HT, Norgaard M. The impact of comorbidity on cancer survival: a review. Clin Epidemiol. 2013 Nov 1;5(Suppl 1):3-29. doi: 10.2147/CLEP.S47150. PMID 24227920
- [Background] Jorgensen TL, Hallas J, Friis S, Herrstedt J. Comorbidity in elderly cancer patients in relation to overall and cancer-specific mortality. Br J Cancer. 2012 Mar 27;106(7):1353-60. doi: 10.1038/bjc.2012.46. Epub 2012 Feb 21. PMID 22353805
- [Background] Sarfati D, Koczwara B, Jackson C. The impact of comorbidity on cancer and its treatment. CA Cancer J Clin. 2016 Jul;66(4):337-50. doi: 10.3322/caac.21342. Epub 2016 Feb 17. PMID 26891458
- [Background] Wedding U, Roehrig B, Klippstein A, Steiner P, Schaeffer T, Pientka L, Hoffken K. Comorbidity in patients with cancer: prevalence and severity measured by cumulative illness rating scale. Crit Rev Oncol Hematol. 2007 Mar;61(3):269-76. doi: 10.1016/j.critrevonc.2006.11.001. Epub 2007 Jan 4. PMID 17207632
- [Background] Abravan A, Faivre-Finn C, Gomes F, van Herk M, Price G. Comorbidity in patients with cancer treated at The Christie. Br J Cancer. 2024 Nov;131(8):1279-1289. doi: 10.1038/s41416-024-02838-w. Epub 2024 Sep 4. PMID 39232185
- [Background] Vrinzen CEJ, Delfgou L, Stadhouders N, Hermens RPMG, Merkx MAW, Bloemendal HJ, Jeurissen PPT. A Systematic Review and Multilevel Regression Analysis Reveals the Comorbidity Prevalence in Cancer. Cancer Res. 2023 Apr 4;83(7):1147-1157. doi: 10.1158/0008-5472.CAN-22-1336. PMID 36779863
- [Background] Siembida EJ, Smith AW, Potosky AL, Graves KD, Jensen RE. Examination of individual and multiple comorbid conditions and health-related quality of life in older cancer survivors. Qual Life Res. 2021 Apr;30(4):1119-1129. doi: 10.1007/s11136-020-02713-0. Epub 2021 Jan 14. PMID 33447956
- [Background] Williams GR, Mackenzie A, Magnuson A, Olin R, Chapman A, Mohile S, Allore H, Somerfield MR, Targia V, Extermann M, Cohen HJ, Hurria A, Holmes H. Comorbidity in older adults with cancer. J Geriatr Oncol. 2016 Jul;7(4):249-57. doi: 10.1016/j.jgo.2015.12.002. Epub 2015 Dec 22. PMID 26725537